CLINICAL TRIAL: NCT03696108
Title: A Phase 3, Randomized, Double-blind Clinical Study to Evaluate the Long-term Safety and Efficacy of MK-7264 in Japanese Adult Participants With Refractory or Unexplained Chronic Cough
Brief Title: A Study of Gefapixant (MK-7264) in Japanese Adult Participants With Refractory or Unexplained Chronic Cough (MK-7264-038)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7264-038; MK-7264-038 (Other: Merck Protocol Number); 184154 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2018-10-03; First posted 2018-10-04 (Actual); Results first posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-08

CONDITIONS: Chronic Cough
MeSH Terms: conditions — Chronic Cough | interventions — Gefapixant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gefapixant 15 mg BID (Experimental): Participants will receive gefapixant 15 mg tablet and placebo tablet to match gefapixant 45 mg twice daily (BID) during the study period (52 weeks).
  Interventions: Drug: Gefapixant; Drug: Placebo
- Gefapixant 45 mg BID (Experimental): Participants will receive gefapixant 45 mg tablet and placebo tablet to match gefapixant 15 mg BID during the study period (52 weeks).
  Interventions: Drug: Gefapixant; Drug: Placebo

INTERVENTIONS:
Drug: Gefapixant — Gefapixant 15 mg or 45 mg tablet administered orally BID
  Other Names: MK-7264
Drug: Placebo — Placebo matched to gefapixant 15 mg or 45 mg administered orally BID

SUMMARY:
The primary objective of this study is to evaluate the safety of two doses of gefapixant (MK-7264) in Japanese adult participants with refractory or unexplained chronic cough.

ELIGIBILITY:
Inclusion Criteria:

* Chest radiograph or computed tomography scan of the thorax not demonstrating any abnormality considered to be significantly contributing to the chronic cough or any other clinically significant lung disease in the opinion of the principal investigator or the sub-investigator.
* Chronic cough for ≥ 4 months and a diagnosis of refractory or unexplained chronic cough.
* Persistent cough, despite treatment in accordance with the latest guideline of cough from the Japanese Respiratory Society, cough is a burden to the participant, and needs further treatment.
* If female, is not pregnant, not breast-feeding, and either is not a woman of childbearing potential or agrees to follow the contraceptive guidance.

Exclusion Criteria:

* Current smoker, or has given up smoking within 12 months of Screening.
* History of upper or lower respiratory tract infection or recent clinically significant change in pulmonary status.
* Has a history of chronic bronchitis.
* Current use of an angiotensin converting enzyme inhibitor (ACEI) or has taken an ACEI within 3 months of Screening.
* Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m^2 OR ≥30 mL/min/1.73 m^2 and <50 mL/min/1.73 m^2 at Visit 1 with unstable renal function (defined as a ≥50% increase of serum creatinine compared to a value obtained at least 6 months prior to Visit 1).
* History of malignancy ≤ 5 years.
* User of recreational or illicit drugs or has had a recent history (within the last year) of drug or alcohol abuse or dependence.
* Systolic blood pressure >160 mm Hg or a diastolic blood pressure >90 mm Hg at Screening.
* History of cutaneous adverse drug reaction to sulfonamide antibiotics or other sulfonamide-containing drugs.
* Known allergy/sensitivity or contraindication to gefapixant.
* Donated or lost ≥1 unit of blood within 8 weeks prior to the first dose of gefapixant.
* Previously received gefapixant or is currently participating in or has participated in an interventional clinical study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (61):
- Japan (61):
  - Chubu Rosai Hospital ( Site 3839), Nagoya, Aichi-ken
  - National Hospital Organization Nagoya Medical Center ( Site 3898), Nagoya, Aichi-ken
  - Nagoya City University Hospital ( Site 3899), Nagoya, Aichi-ken
  - Fukuoka University Chikushi Hospital ( Site 3886), Chikushino-shi, Fukuoka
  - Oishi Clinic ( Site 3818), Kasuya-gun, Fukuoka
  - National Hospital Organization Fukuokahigashi Medical Center ( Site 3849), Koga, Fukuoka
  - Nagata Hospital ( Site 3815), Yanagawa, Fukuoka
  - Tohno Chuo Clinic ( Site 3883), Mizunami, Gifu
  - National Hospital Organization Shibukawa Medical Center ( Site 3843), Shibukawa, Gunma
  - Idaimae Minamiyojo Int Clinic ( Site 3903), Sapporo, Hokkaido
  - Terada Clinic Respiratory Medicine & General Practice ( Site 3907), Himeji, Hyōgo
  - Kinki Central Hospital ( Site 3910), Itami, Hyōgo
  - Kobe City Hospital Organization Kobe City Medical Center West Hospital ( Site 3868), Kobe, Hyōgo
  - National Hospital Organization Mito Medical Center ( Site 3846), Higashiibaraki-gun, Ibaraki
  - National Hospital Organization Ibarakihigashi National Hospital ( Site 3917), Naka-gun, Ibaraki
  - JA Toride Medical Center ( Site 3822), Toride, Ibaraki
  - National Hospital Organization Kasumigaura Medical Center ( Site 3844), Tsuchiura, Ibaraki
  - Ishikawa Prefectural Central Hospital ( Site 3915), Kanazawa, Ishikawa-ken
  - Japan Community Health care Organization Kanazawa Hospital ( Site 3817), Kanazawa, Ishikawa-ken
  - Komatsu Municipal Hospital ( Site 3892), Komatsu, Ishikawa-ken
  - Kamei Internal Medicine and Respiratory Clinic ( Site 3904), Takamatsu, Kagawa-ken
  - Fujisawa City Hospital ( Site 3891), Fujisawa, Kanagawa
  - Association of Healthcare Corporation Koukankai Koukan Clinic ( Site 3878), Kawasaki, Kanagawa
  - Yokohama City Minato Red Cross Hospital ( Site 3906), Yokohama, Kanagawa
  - Saiseikai Yokohamashi Nanbu Hospital ( Site 3897), Yokohama, Kanagawa
  - Kanagawa Cardiovascular and Respiratory Center ( Site 3908), Yokohama, Kanagawa
  - Matsusaka City Hospital ( Site 3825), Matsusaka, Mie-ken
  - Koyama Medical Clinic ( Site 3838), Matsumoto, Nagano
  - Nagaoka Red Cross Hospital ( Site 3877), Nagaoka, Niigata
  - National Hospital Organization Minami-Okayama Medical Center ( Site 3901), Tsukubo-gun, Okayama-ken
  - Kawaguchi Respiratory Clinic ( Site 3890), Higashiosaka, Osaka
  - Kishiwada City Hospital ( Site 3880), Kishiwada, Osaka
  - Sasaki Naika Clinic ( Site 3872), Sakai, Osaka
  - National Hospital Organization Kinki-chuo Chest Medical Center ( Site 3900), Sakai, Osaka
  - Kindai University Hospital ( Site 3871), Sayama, Osaka
  - Sugiura Clinic ( Site 3806), Kawaguchi, Saitama
  - National Hospital Organization Matsue Medical Center ( Site 3848), Matsue, Shimane
  - JapanOrganizationOfOccupationalHealthAndSafety HamamatsuRosaiHospital ( Site 3821), Hamamatsu, Shizuoka
  - Hamamatsu Medical Center ( Site 3866), Hamamatsu, Shizuoka
  - National Hospital Organization Tenryu Hospital ( Site 3823), Hamamatsu, Shizuoka
  - Tokyo Medical University Hachioji Medical Center ( Site 3911), Hachiōji, Tokyo
  - National Hospital Organization Tokyo National Hospital ( Site 3909), Kiyose, Tokyo
  - Kiheibashi Otolaryngology ( Site 3828), Kodaira, Tokyo
  - Shimonoseki City Hospital ( Site 3902), Shimonoseki, Yamaguchi
  - Akita University Hospital ( Site 3851), Akita
  - Fukui-ken Saiseikai Hospital ( Site 3874), Fukui
  - Gifu Prefectural General Medical Center ( Site 3824), Gifu
  - Tochigi Takao Clinic ( Site 3833), Kagoshima
  - Nagano Red Cross Hospital ( Site 3859), Nagano
  - Saiseikai Niigata Hospital ( Site 3831), Niigata
  - Chibana Clinic ( Site 3809), Okinawa
  - Oita Red Cross Hospital ( Site 3837), Ōita
  - Yamagata Clinic ( Site 3813), Ōita
  - Ito ENT Clinic ( Site 3816), Shizuoka
  - Nihonbashi Egawa Clinic ( Site 3805), Tokyo
  - The Fraternity Memorial Hospital ( Site 3873), Tokyo
  - Showa University Hospital ( Site 3896), Tokyo
  - Ebisu Clinic Koukokukai Medical Corporation ( Site 3804), Tokyo
  - Kono Medical Clinic ( Site 3894), Tokyo
  - Medical Corporation Kouwakai Kouwa Clinic ( Site 3895), Tokyo
  - Tokyo Metropolitan Geriatric Hospital ( Site 3905), Tokyo

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Niimi A, Sagara H, Kikuchi M, Arano I, Sato A, Shirakawa M, La Rosa C, Muccino D. A phase 3, randomized, double-blind, clinical study to evaluate the long-term safety and efficacy of gefapixant in Japanese adult participants with refractory or unexplained chronic cough. Allergol Int. 2022 Oct;71(4):498-504. doi: 10.1016/j.alit.2022.05.006. Epub 2022 Jun 23. PMID 35752582

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 175 participants were originally enrolled in the study. 6 participants at one site were excluded from all analyses, including disposition, due to good clinical practice (GCP) noncompliance at the study site.
Groups:
- Gefapixant 15 mg BID: Participants received a gefapixant 15 mg tablet and a placebo tablet to match gefapixant 45 mg twice daily (BID) for 52 weeks
- Gefapixant 45 mg BID: Participants received a gefapixant 45 mg tablet and a placebo tablet to match gefapixant 15 mg BID for 52 weeks
Period: Overall Study
Arm/Group | Gefapixant 15 mg BID | Gefapixant 45 mg BID
Started | 84 | 85
Completed | 80 | 79
Not Completed | 4 | 6
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gefapixant 15 mg BID | Gefapixant 45 mg BID | Total
Number analyzed (Participants) | 84 | 85 | 169
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.2 (14.1) | 57.6 (15.8) | 57.9 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 51 | 106
  Male | 29 | 34 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 84 | 85 | 169
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 84 | 85 | 169
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Time Frame: Up to 54 Weeks
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Gefapixant 15 mg BID: Participants received a gefapixant 15 mg tablet and a placebo tablet to match gefapixant 45 mg BID for 52 weeks
- Gefapixant 45 mg: Participants received a gefapixant 45 mg tablet and a placebo tablet to match gefapixant 15 mg BID for 52 weeks
Arm/Group | Gefapixant 15 mg BID | Gefapixant 45 mg
Number analyzed (Participants) | 84 | 85
Participants | 79 | 82

2. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: as for outcome 1
Time Frame: Up to 52 Weeks
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Gefapixant 15 mg BID | Gefapixant 45 mg
Number analyzed (Participants) | 84 | 85
Participants | 6 | 17

3. Secondary Outcome: Change From Baseline in the Leicester Cough Questionnaire (LCQ) Total Score at Week 12
Description: The LCQ is a 19-item cough-specific health-related quality of life (HRQoL) questionnaire which contains three domains (physical, psychological and social), calculated as a mean score for each domain ranging from 1 to 7 and total score ranging from 3 to 21. Each item on the LCQ is assessed using a 7-point Likert scale ranging from 1 to 7. Higher scores indicate better HRQoL. The least squares mean of the change from baseline is based on a longitudinal analysis of covariance (ANCOVA) model.
Time Frame: Baseline, Week 12
Population: All randomized participants who have taken at least one dose of study treatment and provided at least one baseline and one post-baseline endpoint observations during the treatment period.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Gefapixant 15 mg BID | Gefapixant 45 mg
Number analyzed (Participants) | 84 | 85
Scores on a Scale | 1.4 [0.7 to 2.0] | 0.9 [0.3 to 1.6]

4. Secondary Outcome: Change From Baseline in LCQ Total Score
Description: The LCQ is a 19-item cough-specific HRQoL questionnaire which contains three domains (physical, psychological and social), calculated as a mean score for each domain ranging from 1 to 7 and total score ranging from 3 to 21. Each item on the LCQ is assessed using a 7-point Likert scale ranging from 1 to 7. Higher scores indicate better HRQoL. The least squares mean of the change from baseline is based on a longitudinal analysis of covariance (ANCOVA) model at weeks 4, 8, 12, 24, 38 and 52 of treatment.
Time Frame: Baseline, up to 52 Weeks
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Gefapixant 15 mg BID | Gefapixant 45 mg
Number analyzed (Participants) | 84 | 85
Scores on a Scale
  Week 4 | 0.9 [0.2 to 1.5] | 0.8 [0.2 to 1.4]
  Week 8: number analyzed (Participants) | 83 | 81
  Week 8 | 1.5 [0.8 to 2.1] | 1.2 [0.6 to 1.9]
  Week 12: number analyzed (Participants) | 83 | 81
  Week 12 | 1.4 [0.7 to 2.0] | 0.9 [0.3 to 1.6]
  Week 24: number analyzed (Participants) | 82 | 81
  Week 24 | 1.6 [0.9 to 2.2] | 1.1 [0.4 to 1.8]
  Week 38: number analyzed (Participants) | 82 | 78
  Week 38 | 1.8 [1.1 to 2.4] | 1.2 [0.6 to 1.9]
  Week 52: number analyzed (Participants) | 80 | 79
  Week 52 | 2.3 [1.6 to 2.9] | 1.5 [0.8 to 2.1]

5. Secondary Outcome: Percentage of Participants With a ≥1.3 Point Change From Baseline in the LCQ Total Score
Description: The LCQ is a 19-item cough-specific HRQoL questionnaire which contains three domains (physical, psychological and social), calculated as a mean score for each domain ranging from 1 to 7 and total score ranging from 3 to 21. Each item on the LCQ is assessed using a 7-point Likert scale ranging from 1 to 7. Higher scores indicate better HRQoL. A clinically meaningful improvement from baseline in HRQoL was defined as ≥1.3-point increase in the LCQ total score at weeks 4, 8, 12, 24, 38 and 52 of treatment.
Time Frame: Baseline, Up to 52 Weeks
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Gefapixant 15 mg BID | Gefapixant 45 mg
Number analyzed (Participants) | 84 | 85
Percentage of Participants
  Week 4 | 38.1 | 36.5
  Week 8: number analyzed (Participants) | 83 | 81
  Week 8 | 43.4 | 43.2
  Week 12: number analyzed (Participants) | 83 | 81
  Week 12 | 48.2 | 40.7
  Week 24: number analyzed (Participants) | 82 | 81
  Week 24 | 53.7 | 45.7
  Week 38: number analyzed (Participants) | 82 | 78
  Week 38 | 56.1 | 44.9
  Week 52: number analyzed (Participants) | 80 | 79
  Week 52 | 58.8 | 46.8

ADVERSE EVENTS:
Time Frame: Up to approximately 54 weeks
Description: The all-cause mortality, serious adverse events, and other adverse events population includes all randomized participants who received at least one dose of study treatment, with participants included in the treatment group corresponding to the study treatment they actually received.
Groups:
- Gefapixant 15 mg: Participants received a gefapixant 15 mg tablet and a placebo tablet to match gefapixant 45 mg twice daily (BID) for 52 weeks
Arm/Group | Gefapixant 15 mg | Gefapixant 45 mg
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/85
Serious Adverse Events (participants affected / at risk) | 2/84 | 10/85
Other Adverse Events (participants affected / at risk) | 73/84 | 76/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gefapixant 15 mg (N=84) | Gefapixant 45 mg (N=85)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Embolic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gefapixant 15 mg (N=84) | Gefapixant 45 mg (N=85)
Constipation (Gastrointestinal disorders) | 6 (6) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 5 (5)
Pyrexia (General disorders) | 5 (5) | 6 (7)
Bronchitis (Infections and infestations) | 10 (11) | 3 (3)
Gastroenteritis (Infections and infestations) | 2 (3) | 6 (6)
Nasopharyngitis (Infections and infestations) | 25 (60) | 33 (61)
Pharyngitis (Infections and infestations) | 8 (10) | 4 (6)
Accidental overdose (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Ageusia (Nervous system disorders) | 0 (0) | 5 (5)
Dysgeusia (Nervous system disorders) | 14 (17) | 40 (40)
Headache (Nervous system disorders) | 9 (11) | 3 (3)
Hypogeusia (Nervous system disorders) | 9 (9) | 14 (14)
Taste disorder (Nervous system disorders) | 6 (6) | 10 (10)
Insomnia (Psychiatric disorders) | 1 (1) | 5 (5)
Asthma (Respiratory, thoracic and mediastinal disorders) | 10 (15) | 6 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (34) | 11 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT03696108/Prot_SAP_000.pdf